CLINICAL TRIAL: NCT05188131
Title: Acute Neuroendocrine Response to Intravenous Infusion of Diclofenac Sodium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Ezio Ghigo, Full Professor, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NR-DICLO
Record Dates: First submitted 2021-12-01; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Hypopituitarism
MeSH Terms: conditions — Hypopituitarism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Infusion of Diclofenac Sodium (Experimental): Intravenous Infusion of Diclofenac Sodium in healthy subjects.
  Interventions: Drug: Intravenous Infusion of Diclofenac Sodium
- Intravenous Infusion of Placebo (Placebo Comparator): Intravenous Infusion of Placebo (isotonic saline) in healthy subjects.
  Interventions: Drug: Intravenous Infusion of Placebo

INTERVENTIONS:
Drug: Intravenous Infusion of Diclofenac Sodium — Intravenous Infusion of Diclofenac Sodium is administered at the dose of 75 mg, diluted in 100 ml of isotonic saline, over 15 minutes.
  Arms: Intravenous Infusion of Diclofenac Sodium
Drug: Intravenous Infusion of Placebo — Intravenous Infusion of Placebo (represented by 100 ml of isotonic saline) is administered over 15 minutes.
  Arms: Intravenous Infusion of Placebo

SUMMARY:
The effects of acute administration of non-steroidal anti-inflammatory drugs (NSAIDs) on the neuroendocrine regulation of hydro-electrolytic metabolism are not precisely known to date.

Although the mechanism by which NSAIDs favor the antidiuretic action of vasopressin (AVP) in the kidney has been partially elucidated, their influence on the mechanisms responsible for regulating its secretion are less known. The interactions between NSAIDs and natriuretic peptides are also not entirely certain.

The present pharmacological research study therefore aims to investigate, in a cohort of healthy subjects, the acute effects of intravenous infusion of diclofenac sodium on the neuroendocrine regulation systems of water and salt balance (i.e. the antidiuretic axis and the system of natriuretic peptides).

ELIGIBILITY:
Inclusion Criteria:

- Any adult healthy subject (with age 20-50 years old) not meeting any of the exclusion criteria listed below

Exclusion Criteria:

* BMI < 18.5 kg/m2 or > 25 kg/m2
* Any active pharmacological treatment
* Pregnancy or breastfeeding
* History of polyuria/polydipsia syndrome
* History of dysionia
* History of peptic disease
* History of gastrointestinal bleeding
* History of kidney disease
* History of heart disease
* History of asthma
* Known allergy to NSAIDs
* Any current acute medical condition

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in plasma copeptin levels between baseline and 15 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 15 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 15 minutes from diclofenac/placebo administration.
Change in plasma copeptin levels between baseline and 30 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 30 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 30 minutes from diclofenac/placebo administration.
Change in plasma copeptin levels between baseline and 45 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 45 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 45 minutes from diclofenac/placebo administration.
Change in plasma copeptin levels between baseline and 60 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 60 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 60 minutes from diclofenac/placebo administration.
Change in plasma copeptin levels between baseline and 90 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 90 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 90 minutes from diclofenac/placebo administration.
Change in plasma copeptin levels between baseline and 120 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 120 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 120 minutes from diclofenac/placebo administration.
Change in plasma copeptin levels between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response of the antidiuretic axis to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 15 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 15 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 15 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 30 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 30 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 30 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 45 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 45 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 45 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 60 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 60 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 60 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 90 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 90 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 90 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 120 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 120 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 120 minutes from diclofenac/placebo administration.
Change in plasma MR-proANP levels between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response of the natriuretic peptide system to the administration of intravenous diclofenac sodium, compared to placebo, is evaluated by measuring plasma MR-proANP (pmol/L) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.

SECONDARY OUTCOMES:
Change in serum sodium levels between baseline and 15 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 15 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 15 minutes from diclofenac/placebo administration.
Change in serum sodium levels between baseline and 30 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 30 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 30 minutes from diclofenac/placebo administration.
Change in serum sodium levels between baseline and 45 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 45 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 45 minutes from diclofenac/placebo administration.
Change in serum sodium levels between baseline and 60 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 60 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 60 minutes from diclofenac/placebo administration.
Change in serum sodium levels between baseline and 90 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 90 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 90 minutes from diclofenac/placebo administration.
Change in serum sodium levels between baseline and 120 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 120 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 120 minutes from diclofenac/placebo administration.
Change in serum sodium levels between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 15 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 15 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 15 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 30 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 30 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 30 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 45 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 45 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 45 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 60 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 60 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 60 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 90 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 90 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 90 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 120 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 120 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 120 minutes from diclofenac/placebo administration.
Change in plasma MR-proADM levels between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring plasma MR-proADM (pmol/L) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in urine sodium levels between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring urine sodium (mmol/L) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in urine potassium levels between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring urine potassium (mmol/L) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in urine osmolality between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of glycometabolic and hydroelectrolyte biochemical balance was evaluated by measuring urine osmolality (mOsm/kg) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in resistance at bioimpedance vector analysis between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of bioimpedance vector analysis was evaluated by measuring resistance (Ohm) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in reactance at bioimpedance vector analysis between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of bioimpedance vector analysis (BIVA) was evaluated by measuring reactance (Ohm) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in phase angle at bioimpedance vector analysis between baseline and 240 minutes after diclofenac/placebo administration | From baseline (0 minutes) to 240 minutes after diclofenac/placebo administration
  The response to the administration of intravenous diclofenac sodium, compared to placebo, in terms of bioimpedance vector analysis (BIVA) was evaluated by measuring phase angle (°) at baseline (0 minutes) and after 240 minutes from diclofenac/placebo administration.
Change in late-night salivary cortisol levels between 9 hours before and 15 hours after diclofenac/placebo administration | From 9 hours before to 15 hours after diclofenac/placebo administration
  The influence the administration of intravenous diclofenac sodium, compared to placebo, on late-night salivary cortisol was evaluated by measuring late-night salivary cortisol (ng/ml) at 11 pm the day before diclofenac/placebo administration, and at 11 pm the day of diclofenac/placebo administration.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheung NT, Coley S, Sheeran T, Situnayake RD. Syndrome of inappropriate secretion of antidiuretic hormone induced by diclofenac. BMJ. 1993 Jan 16;306(6871):186. doi: 10.1136/bmj.306.6871.186-a. No abstract available. PMID 8443484
- [Background] Verrua E, Mantovani G, Ferrante E, Noto A, Sala E, Malchiodi E, Iapichino G, Peccoz PB, Spada A. Severe water intoxication secondary to the concomitant intake of non-steroidal anti-inflammatory drugs and desmopressin: a case report and review of the literature. Hormones (Athens). 2013 Jan-Mar;12(1):135-41. doi: 10.1007/BF03401295. PMID 23624139
- [Background] Roche C, Ragot C, Moalic JL, Simon F, Oliver M. Ibuprofen can induce syndrome of inappropriate diuresis in healthy young patients. Case Rep Med. 2013;2013:167267. doi: 10.1155/2013/167267. Epub 2013 Jun 12. PMID 23840216
- [Background] Lim SY, Panikkath R, Prabhakar S. Syndrome of inappropriate antidiuretic hormone secretion associated with prolonged keterolac use. Clin Nephrol Case Stud. 2014 Jan 22;2:5-8. doi: 10.5414/CNCS108083. eCollection 2014. PMID 29043122
- [Background] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Eur J Endocrinol. 2014 Feb 25;170(3):G1-47. doi: 10.1530/EJE-13-1020. Print 2014 Mar. PMID 24569125
- [Background] Murase T, Tian Y, Fang XY, Verbalis JG. Synergistic effects of nitric oxide and prostaglandins on renal escape from vasopressin-induced antidiuresis. Am J Physiol Regul Integr Comp Physiol. 2003 Feb;284(2):R354-62. doi: 10.1152/ajpregu.00065.2002. Epub 2002 Oct 10. PMID 12388460
- [Background] Babina AV, Lavrinenko VA, Shestopalova LV, Ivanova LN. Morphological characteristics of the inner medullary zone in the kidneys of Brattleboro and Wistar rats during blockade of prostaglandin synthesis. Bull Exp Biol Med. 2011 Jun;151(2):268-72. doi: 10.1007/s10517-011-1305-0. PMID 22238766
- [Background] Lavrinenko VA, Babina AV, Shestopalova LV, Beizel NF, Ivanova LN. Effects of sodium diclofenac on the concentration function in animals with different neurohypophyseal status. Bull Exp Biol Med. 2012 Apr;152(6):728-30. doi: 10.1007/s10517-012-1617-8. English, Russian. PMID 22803175
- [Background] Babina AV, Lavrinenko VA. Electron Microscopic Study of the Inner Medulla in Rat Kidneys under Conditions of Vasopressin Treatment Combined with Prostaglandin Synthesis Blockade. Bull Exp Biol Med. 2016 Oct;161(6):850-852. doi: 10.1007/s10517-016-3527-7. Epub 2016 Oct 25. PMID 27783283
- [Background] Lavrinenko VA, Babina AV. Efficiency of Osmotic Concentration after Combined Treatment with Vasopressin and Blockage of Prostaglandin Synthesis. Bull Exp Biol Med. 2016 Dec;162(2):187-190. doi: 10.1007/s10517-016-3572-2. Epub 2016 Dec 2. PMID 27909962
- [Background] Palmer BF, Clegg DJ. Altered Prostaglandin Signaling as a Cause of Thiazide-Induced Hyponatremia. Am J Kidney Dis. 2018 Jun;71(6):769-771. doi: 10.1053/j.ajkd.2017.11.026. Epub 2018 Feb 28. No abstract available. PMID 29501264
- [Background] Puurunen J, Leppaluoto J. Centrally administered PGE2 inhibits gastric secretion in the rat by releasing vasopressin. Eur J Pharmacol. 1984 Sep 3;104(1-2):145-50. doi: 10.1016/0014-2999(84)90381-9. PMID 6094207
- [Background] Bojanowska E, Guzek JW. Inhibition of prostaglandin synthesis and the release of vasopressin and oxytocin from the rat neurohypophysis: in vitro studies. Exp Clin Endocrinol. 1991;98(3):213-21. doi: 10.1055/s-0029-1211120. PMID 1778241
- [Background] Walker BR. Suppressed basal antidiuretic hormone release during cyclooxygenase inhibition in conscious dogs. Am J Physiol. 1983 Apr;244(4):R487-91. doi: 10.1152/ajpregu.1983.244.4.R487. PMID 6404183
- [Background] Heida JE, Boesten LSM, Ettema EM, Muller Kobold AC, Franssen CFM, Gansevoort RT, Zittema D. Comparison of ex vivo stability of copeptin and vasopressin. Clin Chem Lab Med. 2017 Jun 27;55(7):984-992. doi: 10.1515/cclm-2016-0559. PMID 27879483
- [Background] Morgenthaler NG, Struck J, Alonso C, Bergmann A. Assay for the measurement of copeptin, a stable peptide derived from the precursor of vasopressin. Clin Chem. 2006 Jan;52(1):112-9. doi: 10.1373/clinchem.2005.060038. Epub 2005 Nov 3. PMID 16269513
- [Background] Castellani S, Del Rosso A, Chen JL, Camaiti A, Carnovali M, Masotti G. The renal excretory activity of atrial natriuretic factor is independent of renal prostaglandins in humans. Prostaglandins Leukot Essent Fatty Acids. 1991 Jan;42(1):23-9. doi: 10.1016/0952-3278(91)90062-a. PMID 1826370
- [Background] Vlaskovska M, Hertting G, Knepel W. Adrenocorticotropin and beta-endorphin release from rat adenohypophysis in vitro: inhibition by prostaglandin E2 formed locally in response to vasopressin and corticotropin-releasing factor. Endocrinology. 1984 Sep;115(3):895-903. doi: 10.1210/endo-115-3-895. PMID 6204854
- [Background] Okajima T, Heldt R, Hertting G. Functional compartmentalization of arginine-vasopressin-activated cyclic AMP in anterior pituitary gland: the presence of a compartment activated by prostaglandin E2. Life Sci. 1986 Mar 24;38(12):1143-9. doi: 10.1016/0024-3205(86)90251-1. PMID 3007904
- [Background] Thompson ME, Hedge GA. Inhibition of corticotropin secretion by hypothalamic administration of indomethacin. Neuroendocrinology. 1978;25(4):212-20. doi: 10.1159/000122743. PMID 206852
- [Background] Lukaski HC, Vega Diaz N, Talluri A, Nescolarde L. Classification of Hydration in Clinical Conditions: Indirect and Direct Approaches Using Bioimpedance. Nutrients. 2019 Apr 10;11(4):809. doi: 10.3390/nu11040809. PMID 30974817